CLINICAL TRIAL: NCT00712959
Title: Immune Responses in Adults to Revaccination With Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (ADACEL®) 10 Years After a Previous Dose
Brief Title: Immune Responses in Adults to Revaccination With ADACEL® 10 Years After a Previous Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TD526
Record Dates: First submitted 2008-07-07; First posted 2008-07-10 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Pertussis; Tetanus; Diphtheria
Keywords: Pertussis; Tetanus; Diphtheria; Acellular pertussis; ADACEL®,; Tdap vaccine
MeSH Terms: conditions — Whooping Cough; Tetanus; Diphtheria | interventions — Tetanus Toxoid; adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Previous Tdap or Tdap-IPV Recipients (Experimental): Participants received Tdap or Tdap-Inactivated Poliomyelitis Vaccine (IPV) in a previous study (TD9707 or TD9805)
  Interventions: Biological: Tetanus, Reduced Diphtheria Toxoid and Acellular Pertussis (ADACEL®)
- Group 2: Tdap vaccine-naïve (Active Comparator): Participants are age-balanced Tdap vaccine-naïve and will receive Tdap vaccine in the study at least 10 years after a previous tetanus, diphtheria and/or pertussis dose.
  Interventions: Biological: Tetanus, Reduced Diphtheria Toxoid and Acellular Pertussis (ADACEL®)
- Group 3 (No Intervention): Past participants in Study TD9707 and TD9805 did not qualify for Tdap re-administration in this study or were unwilling to receive a second dose of Tdap. They were not included in the analysis for the study

INTERVENTIONS:
Biological: Tetanus, Reduced Diphtheria Toxoid and Acellular Pertussis (ADACEL®) — 0.5 ml, IM
  Other Names: Tdap; ADACEL®
  Arms: Group 1: Previous Tdap or Tdap-IPV Recipients
Biological: Tetanus, Reduced Diphtheria Toxoid and Acellular Pertussis (ADACEL®) — 0.5 mL, IM
  Other Names: Tdap; Adacel®
  Arms: Group 2: Tdap vaccine-naïve

SUMMARY:
The purpose of this study is to collect additional immunogenicity and safety data on re-dosing with Tdap vaccine (ADACEL®) in a continuing effort to address the public health need to establish broader population immunity against pertussis, as well as diphtheria and tetanus.

Primary Objective:

* To assess immune response to Tdap vaccine (ADACEL®) one month after booster vaccination.

DETAILED DESCRIPTION:
This is an open-label, multicenter study to describe the immunological response and safety of repeat administration of an adolescent/adult-formulation tetanus-diphtheria-acellular pertussis Tdap vaccine (ADACEL®), 10 years following initial administration of Tdap vaccine.

ELIGIBILITY:
Inclusion Criteria :

* Received Tdap or Tdap-IPV vaccine in study TD9707 or TD9805.
* Never previously received Tdap vaccine and has not received any tetanus-, diphtheria , or pertussis-containing vaccine in the past 10 years.
* Participated in TD9707 or TD9805 but does not meet inclusion/ exclusion criteria or willing to undergo phlebotomy but not willing to receive Tdap (ADACEL®) vaccine.
* Signed Institutional Review Board (IRB)-approved informed consent form
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman, a negative urine pregnancy test and the use of effective method(s) of contraception, or the inability to become pregnant

Exclusion Criteria :

* Any condition listed as a contraindication in the ADACEL® Canadian product monograph
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine
* Chronic illness, at a stage that could interfere with trial conduct or completion, in the opinion of the investigator
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic (injected or oral) corticosteroid therapy. Individuals on a tapering dose schedule of oral steroids lasting less than 7 days may be included in the trial as long as they have not received more than 1 course within the last 2 weeks prior to enrollment
* Febrile illness (temperature ≥ 37.5°C [99.5°F]) at the time of inclusion
* History of documented diphtheria, pertussis, or tetanus disease since participation in studies TD9707 or TD9805. Or history of documented diphtheria, pertussis, or tetanus disease in the last 10 years.
* Known or suspected receipt of a diphtheria-, pertussis-, or tetanus-containing vaccine since participation in study TD9707 or TD9805. For Group 2, known or suspected receipt of a diphtheria-, pertussis-, or tetanus-containing vaccine in the last 10 years.
* Receipt of any vaccine, other than influenza vaccine, in the 28-day period prior to Visit 1 or scheduled to receive any vaccine, other than influenza vaccine, in the period between Visit 1 and Visit 2. For influenza vaccine only, defer if received in the 14 days prior to enrollment or scheduled to receive prior to Visit 2.
* Receipt of blood or blood-derived products in the past 3 months
* Suspected or known hypersensitivity to any of the vaccine components, or a life-threatening reaction after previous administration of the vaccine or a vaccine containing the same substances
* Unable to attend the scheduled visits or to comply with the study procedures
* In females of childbearing potential, known pregnancy or positive serum/urine pregnancy test
* Breast-feeding woman
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding enrollment. Planned participation in another clinical trial during the present trial period
* Current alcohol or recreational drug use that may interfere with the subject's ability to comply with trial procedures
* Thrombocytopenia, bleeding disorder, anticoagulation therapy contraindicating intramuscular (IM) vaccination
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* Other events which in the judgment of the investigator would preclude vaccination at the time of Visit 1 For Group 3
* History of documented diphtheria, pertussis, or tetanus disease since participation in study TD9707 or TD9805
* Known or suspected receipt of a diphtheria-, pertussis-, or tetanus-containing vaccine since participation in study TD9707 or TD9805.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 769 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (7):
- Canada (7):
  - Coquitlam, British Columbia
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Pierrefonds, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec

REFERENCES:
- [Result] Halperin SA, Scheifele D, De Serres G, Noya F, Meekison W, Zickler P, Larrivee L, Langley JM, McNeil SA, Dobson S, Jordanov E, Thakur M, Decker MD, Johnson DR. Immune responses in adults to revaccination with a tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine 10 years after a previous dose. Vaccine. 2012 Jan 20;30(5):974-82. doi: 10.1016/j.vaccine.2011.11.035. Epub 2011 Nov 21. PMID 22115634
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 26 June 2008 to 27 February 2009 at 7 medical centers in Canada.
Pre-assignment Details: A total of 769 participants who met the inclusion and exclusion criteria were enrolled, 768 were vaccinated and evaluated.
Groups:
- Group 2: Tdap Vaccine-naïve: Age-balanced Tdap vaccine-naïve participants who received Tdap vaccine in the study at least 10 years after a previous tetanus, diphtheria and/or pertussis dose.
Period: Overall Study
Arm/Group | Group 1: Previous Tdap or Tdap-IPV Recipients | Group 2: Tdap Vaccine-naïve
Started | 361 | 407
Completed | 342 | 404
Not Completed | 19 | 3
Not completed — Protocol Violation | 3 | 1
Not completed — Lost to Follow-up | 13 | 2
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Previous Tdap or Tdap-IPV Recipients: Participants received Tdap or Tdap-IPV in a previous study (TD9707 or TD9805)
- Total: Total of all reporting groups
Arm/Group | Group 1: Previous Tdap or Tdap-IPV Recipients | Group 2: Tdap Vaccine-naïve | Total
Number analyzed (Participants) | 361 | 407 | 768
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 356 | 402 | 758
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.2 (14.0) | 34.6 (12.5) | 33.0 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 264 | 458
  Male | 167 | 143 | 310
Region of Enrollment [Number; unit: participants]
  Canada | 361 | 407 | 768

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroprotection Against Tetanus and Diphtheria Before and After Revaccination With ADACEL® 10 Years After a Previous Dose
Description: Diphtheria concentrations were determined by neutralization assay; tetanus concentrations were determined by enzyme-linked immunosorbent assay (ELISA).
  Seroprotection was defined as anti-tetanus or anti-diphtheria concentrations ≥ 0.1 IU/mL.
Time Frame: Day 0 (pre-vaccination) and 30 post-vaccination
Population: Anti-tetanus and anti-diphtheria concentrations were assessed in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Previous Tdap or Tdap-IPV Recipients | Group 2: Tdap Vaccine-naïve
Number analyzed (Participants) | 324 | 381
Percentage of Participants
  Anti-tetanus Pre-vaccination | 45 | 49
  Anti-tetanus Post-vaccination | 100 | 100
  Anti-Diphtheria Pre-vaccination | 74 | 66
  Anti-Diphtheria Post-vaccination | 99 | 96

2. Primary Outcome: Anti-Pertussis Geometric Mean Concentrations Post-vaccination With ADACEL® 10 Years After a Previous Dose
Description: Post-vaccination geometric mean concentrations (GMCs) for pertussis toxoid (PT), filamentous hemagglutinin (FHA), pertactin (PRN), and fimbriae types 2 and 3 (FIM), were determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 30 post-vaccination
Population: Geometric mean concentrations were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: Previous Tdap or Tdap-IPV Recipients | Group 2: Tdap Vaccine-naïve
Number analyzed (Participants) | 324 | 381
EU/mL
  Pertussis Toxoid [n=318, 357] | 116 [105 to 129] | 89.2 [80.2 to 99.3]
  Filamentous Haemagglutinin [n=324, 380] | 214 [199 to 231] | 249 [229 to 272]
  Pertactin [n=324, 381] | 266 [243 to 292] | 216 [188 to 247]
  Fimbriae Types 2 and 3 [n=324, 378] | 779 [720 to 843] | 1015 [894 to 1154]

3. Other Pre Specified Outcome: Percentage of Participants Achieving Booster Response of Anti-Tetanus and Anti-Diptheria Following Revaccination With ADACEL® 10 Years After a Previous Dose
Description: Anti-diphtheria or anti-tetanus booster responses were defined as:
  Pre-vaccination antibody concentrations of < 0.1 IU/mL and a post-vaccination levels ≥ 0.4 IU/mL; or a pre-vaccination antibody concentrations of ≥ 0.1 IU/mL to < 2 IU/mL and a 4-fold rise; or pre-vaccination antibody concentrations of ≥ 2.0 IU/mL and a 2-fold response.
Time Frame: Day 30 post-vaccination
Population: Booster Response to Tetanus and Diptheria antigens were assessed in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Previous Tdap or Tdap-IPV Recipients | Group 2: Tdap Vaccine-naïve
Number analyzed (Participants) | 324 | 381
Percentage of Participants
  Anti-Tetanus [N = 324, 379] | 83 | 82
  Anti-Diphtheria [N = 324, 381] | 86 | 81

4. Other Pre Specified Outcome: Percentage of Participants Achieving Booster Response for Each Anti-Pertussis Antibody Following Revaccination With ADACEL® 10 Years After a Previous Dose
Description: Booster response for each anti-pertussis antibody was defined as a post-vaccination antibody concentration:
  * ≥ 4 x the Lower limit of quantitation (LLOQ), if the pre-vaccination concentration was < LLOQ; or
  * ≥ 4 x the pre-vaccination antibody concentration, if the pre-vaccination concentration was ≥ LLOQ but < 4 x LLOQ; or
  * ≥ 2 x the pre-vaccination antibody concentration, if the pre-vaccination concentration was ≥ 4 x LLOQ.
Time Frame: Day 30 post-vaccination
Population: Booster response for each anti-Pertussis antibody was assessed in the per-protocol population.
Measure: Number; unit: Percentage of Particpants
Arm/Group | Group 1: Previous Tdap or Tdap-IPV Recipients | Group 2: Tdap Vaccine-naïve
Number analyzed (Participants) | 324 | 381
Percentage of Particpants
  Anti-Pertussis Toxoid [N = 285, 330] | 88 | 84
  Filamentous Haemagglutinin [N = 324, 379] | 88 | 94
  Pertactin [N = 324, 381] | 90 | 93
  Fimbriae Types 2 and 3 [N = 324, 371] | 84 | 93

5. Other Pre Specified Outcome: Geometric Mean Concentrations Against Pertussis Antigens Before and Post-vaccination With ADACEL® 10 Years After a Previous Dose
Description: Post-vaccination geometric mean concentrations (GMCs) against pertussis toxoid (PT), filamentous hemagglutinin (FHA), pertactin (PRN), and fimbriae types 2 and 3 (FIM), were determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 0 (pre-vaccination) and Day 30 post-vaccination
Population: Geometric mean concentrations were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: Previous Tdap or Tdap-IPV Recipients | Group 2: Tdap Vaccine-naïve
Number analyzed (Participants) | 324 | 381
EU/mL
  Pertussis Toxoid [Pre, N = 291, 353] | 15.1 [12.9 to 17.6] | 9.42 [8.20 to 10.8]
  Pertussis Toxoid [Post, N = 318, 357] | 116 [105 to 129] | 89.2 [80.2 to 99.3]
  Filamentous Haemagglutinin [Pre, N = 324, 380] | 34.8 [31.2 to 38.7] | 20.0 [17.7 to 22.5]
  Filamentous Haemagglutinin [Post, N = 324, 380] | 214 [199 to 231] | 249 [229 to 272]
  Pertactin [Pre, N = 324, 381] | 28.2 [24.4 to 32.7] | 8.54 [7.41 to 9.85]
  Pertactin [Post, N = 324, 381] | 266 [243 to 292] | 216 [188 to 247]
  Fimbriae Types 2 and 3 [Pre, N = 324, 374] | 124 [111 to 139] | 37.8 [32.7 to 43.7]
  Fimbriae Types 2 and 3 [Post, N=324, 378] | 779 [720 to 843] | 1015 [894 to 1154]

6. Other Pre Specified Outcome: Geometric Mean Concentrations Against Tetanus and Diphtheria Antigens Before and Post-vaccination With ADACEL® 10 Years After a Previous Dose
Description: Post-vaccination geometric mean concentrations (GMCs) for Diphtheria was determined by neutralization assay; GMCs for tetanus was determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 0 (pre-vaccination) and Day 30 post-vaccination
Population: Geometric mean concentrations were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group 1: Previous Tdap or Tdap-IPV Recipients | Group 2: Tdap Vaccine-naïve
Number analyzed (Participants) | 324 | 381
IU/mL
  Anti-Tetanus [Pre, N = 324, 379] | 0.835 [0.754 to 0.924] | 0.778 [0.679 to 0.892]
  Anti-Tetanus [Post, N = 324, 381] | 8.79 [8.06 to 9.59] | 9.64 [8.73 to 10.7]
  Anti-Diphtheria [Pre, N = 324, 381] | 0.283 [0.235 to 0.341] | 0.198 [0.163 to 0.240]
  Anti-Diphtheria [Post, N = 324, 381] | 4.06 [3.49 to 4.71] | 2.74 [2.36 to 3.18]

7. Other Pre Specified Outcome: Number of Participants Reporting at Least One Solicited Injection Site or Systemic Reaction Post-vaccination With ADACEL® 10 Years After a Previous Dose
Description: Solicited Injection Site Reactions: Pain, Erythema, and swelling. Solicited Systemic Reactions: Fever (temperature), Headache, Malaise, and Myalgia.
  Grade 3 - Pain: Incapacitating, : Incapacitating, unable to perform usual activities, may have/or required medical care or absenteeism; Erythema and Swelling: ≥5 cm; Fever: > 39.0°C, Headache, Malaise, and Myalgia Prevents daily activities.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Group 1: Previous Tdap or Tdap-IPV Recipients | Group 2: Tdap Vaccine-naïve
Number analyzed (Participants) | 361 | 407
Participants
  Any Pain [N = 352, 404] | 309 | 341
  Grade 3 Pain [N = 352, 404] | 9 | 7
  Any Erythema [N = 351, 404] | 81 | 120
  Grade 3 Erythema [N = 351, 404] | 7 | 7
  Any Swelling [N= 352, 403] | 72 | 94
  Grade 3 Swelling [N= 352, 403] | 9 | 7
  Any Fever [N = 356, 405] | 15 | 20
  Grade 3 Fever [N = 356, 405] | 0 | 0
  Any Headache [N = 350, 404] | 142 | 152
  Grade 3 Headache [N = 350, 404] | 6 | 8
  Any Malaise [N = 350, 404] | 103 | 117
  Grade 3 Malaise [N = 350, 404] | 7 | 8
  Any Myalgia [N = 351, 404] | 211 | 216
  Grade 3 Myalgia [N = 351, 404] | 8 | 6

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 (post-vaccination) up to 6 months post-vaccination
Description: The diary cards for solicited safety data were not returned for some participants; the total number for each event therefore represents those with available data for the indicated event.
Arm/Group | Group 1: Previous Tdap or Tdap-IPV Recipients | Group 2: Tdap Vaccine-naïve
Serious Adverse Events (participants affected / at risk) | 3/361 | 1/407
Other Adverse Events (participants affected / at risk) | 309/361 | 341/407
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Previous Tdap or Tdap-IPV Recipients (N=361) | Group 2: Tdap Vaccine-naïve (N=407)
Arnold-Chiari Malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaginal Haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: Previous Tdap or Tdap-IPV Recipients (N=361) | Group 2: Tdap Vaccine-naïve (N=407)
Solicited Injection Site Pain (General disorders) | 309/352 (309) | 341/404 (341)
Solicited Injection Site Erythema (General disorders) | 81/351 (81) | 120/404 (120)
Malaise (General disorders) | 103/350 (103) | 117/404 (117)
Solicited Injection Site Swelling (General disorders) | 72/351 (72) | 94/403 (94)
Myalgia (Musculoskeletal and connective tissue disorders) | 211/351 (211) | 216/404 (216)
Headache (Nervous system disorders) | 142/350 (142) | 152/404 (152)
Headache (Nervous system disorders) | 13 (13) | 36 (36)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 22 (23)
Nasopharyngitis (Infections and infestations) | 30 (31) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications